CLINICAL TRIAL: NCT01394354
Title: Safety of Vorinostat in Combination With Bortezomib, Doxorubicin and Dexamethasone (VBDD) in Patients With Refractory or Relapsed Multiple Myeloma, A Phase I/II Study, Short Title: VBDD
Brief Title: Vorinostat in Combination With Bortezomib, Doxorubicin and Dexamethasone (VBDD) in Patients With Refractory or Relapsed Multiple Myeloma (MM)
Acronym: VBDD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Janssen-Cilag Ltd. (Industry)
Responsible Party: Principal Investigator, Monika Engelhardt, Prof. Dr. med., University Hospital Freiburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00658, MK-0683-201
Record Dates: First submitted 2011-06-21; First posted 2011-07-14 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Multiple Myeloma in Relapse
Keywords: Multiple Myeloma relapsed refractory
MeSH Terms: interventions — Vorinostat; Bortezomib; Doxorubicin; Dexamethasone; dexamethasone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Vorinostat. To determine the MTD, dose escalation for Vorinostat will be conducted following the "3 + 3 design The first cohort of 3 patients will be given 100mg/d on days 1-4, 8-11, 15-18. The second cohort of 3 new patients will be treated with Vorinostat 200mg/d. The third cohort will be given Vorinostat 300mg/d. Cycles will be repeated every 28 days. Maximum treatment cycles: 6. Bortezomib will be administered intravenously (i.v.) 1.3mg/m2 BSA an days 1, 8, 15.
  Doxorubicin will be administered i.v. with a total dose of 18mg/m2 BSA per cycle (9mg/m2 BSA, d1 and 8).
  Dexamethasone will be administered per os (p.o.) with 40mg (first cycle) or 20mg (all other cycles) on d1, 8, 15, and 22.
  Interventions: Drug: Vorinostat; Drug: Bortezomib; Drug: Doxorubicin; Drug: Dexamethasone

INTERVENTIONS:
Drug: Vorinostat — Vorinostat 100 mg/d p.o., on day 1-4, 8-11, and 15-18 /28 day treatment cycle in combination with BDD.
  The dose level of Vorinostat will be escalated in each new cohort:
  if no dose limiting toxicity (DLT) has been observed in the previous dose level in 3 patient, the second cohort of 3 new patients will be treated with Vorinostat 200 mg/d p.o. and the third cohort will be given Vorinostat with 300 mg/d p.o.
  Other Names: ZOLINZA®, ATC code: L01XX
Drug: Bortezomib — 1.3mg/m2 (days 1,8,15)/28 day treatment cycle, i.v., for max. 6 treatment cycles
  Other Names: VELCADE®, ATC code: L01XX32
Drug: Doxorubicin — 18mg/m2 i.v. (days 1 and 8)/ 28 day treatment cycle, max. 6 treatment cycles
  Other Names: ADRIMEDAC®
Drug: Dexamethasone — 40mg abs. p.o. (days 1,8,15,22) 1st treatment cycle, 20mg abs. p.o.(days 1,8,15,22) 2-6 treatment cycles
  Other Names: FORTECORTIN®

SUMMARY:
Primary objective of the study is the determination of the maximum tolerated dose (MTD) of Vorinostat (V), given in combination with fixed doses of Doxorubicin (D), Bortezomib (B) and Dexamethasone (D).

Secondary objectives are:

Assessment of safety and tolerability of VBDD; efficacy data of VBDD.

DETAILED DESCRIPTION:
A first cohort of three patients will be treated at the starting dose level of Vorinostat 100 mg/d, on day 1-4, 8-11, and 15-18 in combination with BDD.

The dose level of Vorinostat will be escalated in each new cohort:

if no dose limiting toxicity (DLT) has been observed in the previous dose level in 3 patient, the second cohort of 3 new patients will be treated with Vorinostat 200 mg/d and the third cohort will be given Vorinostat with 300 mg/d.

Bortezomib will be administered intravenously (i.v.) 1.3mg/m2 d1, 8, 15. Doxorubicin will be administered i.v. with a total dose of 18 mg/m2 per cycle (9 mg/m2, d1 and 8).

Dexamethasone will be administered per os (p.o.) with 40mg (first cycle) and 20mg (all other subsequent cycles) on d1, 8, 15, 22.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory or relapsed MM after at least first-line chemotherapy (CTx) or PBSCT (autologous and allogeneic SCT). All lines of relapse are eligible.
* KPS ≥60%
* Adequate BM function
* Adequate hepatic and renal function (AST and ALT ≤2.5 times ULN, Bilirubin ≤1.5 times ULN, eGFR >20 ml/min)

Exclusion Criteria:

* Patient has had prior treatment with Vorinostat or HDAC inhibitors
* Patients with severe hepatic impairment or acute diffuse infiltrative pulmonary and pericardial disease
* Patient has preexisting NCI CTC ≥grade 3 neuropathy
* Patient with known CNS MM-involvement and/or MM-related/induced meningitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Maximal Tolerated Dose (MTD) | 28 days (within first treatment cycle)
  The Maximal Tolerated Dose (MTD) is estimated as the highest dose at which less than two DLTs in 6 patients are observed in the first cycle. MTD estimation is based on the phase I part of the trial. However, the number of DLT's in the first cycle of the phase II patients will be inspected and discussed as well. The primary target variable is the occurrence of any dose-limiting toxicity (DLT) in MM patients during the first 28 days of treatment.

SECONDARY OUTCOMES:
Response | up to 1 year after inclusion of the last patient
  complete remission (CR, including stringent CR [sCR]), very good partial response (vgPR), partial remission (PR), stable disease (SD), progressive disease (PD). These parameters will be evaluated according to IMWG criteria.
Rates of Adverse Events (AE),Serious Adverse Events and AEs leading to permanent treatment discontinuation | 9 months
  throughout time of treatment (6 months) + 3 months after end of treatment (Follow-up).
  Rates of AE, Serious AE and AEs leading to permanent treatment discontinuation will be provided with accompanying 2-sided 95% confidence intervals. Safety parameters will be analyzed descriptively.
  An AE is any untoward medical occurrence in a patient administered any dose of VBDD study drugs and is defined in detail in the clinical trial protocol. An AE can be any unfavorable sign (incl. an abnormal lab and ECG-findings etc.), symptom, or disease related or not to the study drug.
Quality of Life | during screening period (within 28 days) before start of treatment and at EOT (whether after the completion of the anticipated 6 cycles of chemotherapy or at an earlier time point if patient has to stop treatment because of clinical reasons)
  Assessment with Quality of Life-Questionnaire SF-12
Duration of Response | up to one year after inclusion of the last patient
  Clinical assessment
Progression-free survival (PFS) | up to 1 year after inclusion of the last patient
  estimation by using Kaplan-Meier method
Overall survival (OS) | up to 1 year after inclusion of the last patient
  estimation by using Kaplan-Meier method

CONTACTS AND LOCATIONS:
Overall Officials: Monika Engelhardt, MD, Principal Investigator — University of Freiburg Medical School
Locations (1):
- University Medical Center Freiburg, Freiburg im Breisgau, Germany